CLINICAL TRIAL: NCT04178252
Title: Effectiveness of Eye Mask and Noise Reduction Headset in Emergency Treatment of Primary Headache
Brief Title: Effectiveness of Eye Mask and Headset in Primary Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gul Pamukcu Gunaydin, MD, Faculty Member of Ankara Yildirim Beyazıt University, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AYBU1
Record Dates: First submitted 2019-10-08; First posted 2019-11-26 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Primary Headache Disorder
MeSH Terms: conditions — Headache Disorders, Primary | interventions — Masks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- standard drug (Active Comparator): Standard treatment of primary headache with 10 mg metoclopramide IV in 150 ml saline given over 10 minutes
  Interventions: Other: standard drug
- drug mask (Active Comparator): Standard treatment plus eye mask
  Interventions: Other: mask; Other: standard drug
- drug headset (Active Comparator): Standard treatment plus headset
  Interventions: Other: headset; Other: standard drug
- drug mask headset (Active Comparator): Standard treatment plus headset plus eye mask
  Interventions: Other: mask; Other: headset; Other: standard drug

INTERVENTIONS:
Other: mask — investigators will add eye mask to standard treatment
  Arms: drug mask; drug mask headset
Other: headset — investigators will add headset to standard treatment
  Arms: drug headset; drug mask headset
Other: standard drug — investigators will use 10 mg metoclopramide in 150 ml saline given IV over 10 minutes

SUMMARY:
Primary headache can be triggered by light or noise. Getting rest in a quiet and dark environment for the treatment of acute headache is recommended for relief of pain during an attack. It is hard to provide this kind of environment in a busy emergency department. We aimed to determine if eye masks and noise reduction head sets are effective in reducing pain scores, fastening pain relief when used together with standard care. We also aimed to see if these methods were preferred over standard care.

ELIGIBILITY:
Inclusion Criteria:

* patients with current headache as a chief complaint presenting to Emergency Department
* triage category 3,4,5.
* preliminary clinical diagnosis of primary headache is made after brief history and physical exam by the attending emergency physician according to International Classification of Headache disorders version 3
* the attending physician ordered IV treatment

Exclusion Criteria:

* pregnant
* known or suspected diagnosis of a secondary etiology of headache at presentation or at any point during the Emergency Department visit
* head trauma within 14 days
* inability comply with the study due to insufficient knowledge of Turkish language
* known allergy to standard treatment or rescue treatment
* history of GI bleeding in the last year
* taking any analgesic drug in the last four hours or taking the maximum dose of standard treatment before coming to Emergency Department
* hepatic or renal failure
* patients with hearing or vision loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
change in pain | 30 min
  Change in pain measured by visual analogue scale from baseline measurement achieved at min 0. Investigators will use a 100mm visual analogue scale in which 0 represents no pain and 100 mm represents worse pain ever
change in pain | 60 min
  Change in pain measured by visual analogue scale from baseline measurement achieved at min 0. Investigators will use a 100mm visual analogue scale in which 0 represents no pain and 100 mm represents worse pain ever

SECONDARY OUTCOMES:
need for rescue analgesic drug | 60 min
  Patients will be asked in one question if they need any additional analgesic or if they are comfortable enough. If a patients wants additional analgesics, regardless of their pain score measured by Visual analogue scale he/she will be given dexketoprofen
preference of method over standard treatment | 60 min
  Patients will be asked in one question if they will prefer the method of treatment that they received in the study in case they have headache in the future

CONTACTS AND LOCATIONS:
Overall Officials: Gül Pamukçu Günaydın, MD, Principal Investigator — Ankara Yildirim Beyazit University Faculty of Medicine
Locations (1):
- AnkaraCHBilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anagnostou E, Vikelis M, Tzavellas E, Ghika A, Kouzi I, Evdokimidis I, Kararizou E. Photophobia in primary headaches, in essential blepharospasm and in major depression. Int J Neurosci. 2017 Aug;127(8):673-679. doi: 10.1080/00207454.2016.1231185. Epub 2016 Sep 13. PMID 27580344
- [Background] Wang J, Huang Q, Li N, Tan G, Chen L, Zhou J. Triggers of migraine and tension-type headache in China: a clinic-based survey. Eur J Neurol. 2013 Apr;20(4):689-96. doi: 10.1111/ene.12039. Epub 2013 Jan 28. PMID 23356519
- [Background] Oktay C, Eken C, Goksu E, Dora B. Contribution of verbal suggestion to the therapeutic efficacy of an analgesic agent for acute primary headache. Cephalalgia. 2015 Jun;35(7):579-84. doi: 10.1177/0333102414553821. Epub 2014 Oct 10. PMID 25304763
- [Derived] Pamukcu Gunaydin G, Yildirim C, Sener A, Hassanien NTF. Earmuff and eye mask in the treatment of acute primary headache in emergency department: a randomized controlled open label study. BMC Emerg Med. 2025 Nov 28;25(1):249. doi: 10.1186/s12873-025-01405-7. PMID 41315996